CLINICAL TRIAL: NCT04008433
Title: Median Effective Dose of Lidocaine for the Prevention of Pain Caused by the Injection of Propofol Formulated With Medium-/Long-chain Triglycerides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Director, Yangzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20190604
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Lidocaine; Injection Pain
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lidocaine pre-intravenous injection (Experimental): The initial dose of lidocaine for pre-injection was set at 0.5mg /kg according to previous literature and preliminary test results. The dose of lidocaine was according to the patients' pain level. If there is no pain (negative reaction), the dose of lidocaine in the next patient will be reduced until the patient has pain. If there is pain (positive reaction), the dose of lidocaine will be increased in the next patient until the patient is painless.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Advanced intravenous injection of lidocaine before the propofol injection

SUMMARY:
Propofol is widely used in general anesthesia induction, but the occurrence of peripheral intravenous pain is relatively high, causing anxiety, fear and other adverse emotions in patients , aggravating the stress response, and even leading to adverse events of cardiovascular system . The use of mediate-long chain fat emulsion propofol partly reduces the incidence of injection pain but patients can still suffer from different degrees of pain. Advanced intravenous injection of lidocaine can alleviate the pain of propofol injection, but its application method and dose are controversial. It is worthy of further discussion on how to select the appropriate dose of advanced intravenous injection of lidocaine to effectively prevent the injection pain of mediate-long chain fat emulsion propofol, and simultaneously avoid the adverse reactions of intravenous lidocaine, thus improving patient satisfaction and perioperative safety. In this study, in order to provide clinical references, sequential method was used to find the median effective dose (ED50) by means of pre-intravenous injection of lidocaine to suppress pain in mediate-long chain fat emulsion propofol injection.

ELIGIBILITY:
Inclusion Criteria:

* Ages ranged from 18 to 65.
* ASA Ⅰ or Ⅱ level.

Exclusion Criteria:

* Allergy or contraindication to lidocaine or propofol; required for Central venipuncture catheterization;
* Abnormal liver or kidney function;
* Heavy drinking and long-term use of sedatives, analgesics or anti-anxiety drugs;
* Hearing and language impairment;
* Peripheral vascular disease;
* Severe cardiovascular disease or neurological disorders;
* Failure of one-time peripheral venipuncture;
* Infection of hand or wrist skin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
The appearance of intravenous injection pain | through study completion, an average of 2 minutes
  Yes or No

SECONDARY OUTCOMES:
The levels of intravenous injection pain | through study completion, an average of 2 minutes
  The intravenous injection pain in this study was divided into the following 5 levels according to its severity: level 0: After repeated questioning, the patient did not feel any abnormal sensation; level 1: upon inquiry, the patient felt swelling at the intravenous injection site; Level 2: Upon inquiry, the patient felt pain and had no body movement reaction (facial pain expression, arm withdrawal, tears, etc.); Level 3: Upon inquiry, the patient had pain and body movement reaction. Or complain of pain without inquiry; Level 4: the patient has a strong reaction and body movement reaction. Level 2 and above is defined as injection pain.
If any adverse memory or pain during the induction of general anesthesia | Before patients left the postanesthetic care unit (PACU)
  Patients recalled by visual analogue scale (VAS) to assess injection pain level : Mark 0 is painless. Mark 10 is violent pain, The numbers between them was pain of varying degrees.

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou, Jiangsu, China